CLINICAL TRIAL: NCT01415934
Title: Multisite Randomized Controlled Trial of Continuing vs. Discontinuing Statins
Brief Title: Statin Discontinuation in Advanced Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-0314; UC4NR012584 (NIH)
Record Dates: First submitted 2011-05-10; First posted 2011-08-12 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Palliative Medicine; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continue Statins (No Intervention): Participant will continue on statins as per usual
- Discontinue statins (Experimental): Participant will stop taking their statin drugs
  Interventions: Other: discontinue statins

INTERVENTIONS:
Other: discontinue statins — patients will be randomized to either continue taking statins or discontinue.
  Arms: Discontinue statins

SUMMARY:
The purpose of this study is to determine if there is a difference in survival rate at 60 days after enrollment between patients with advanced life-limiting illness for whom statins are discontinued vs. for patients with advanced life-limiting illness who are maintained on the medication. Secondary outcomes of this study will determine the effects of medication cessation on overall survival, important cardiovascular events, quality of life (QOL), symptoms, performance status, polypharmacy issues, satisfaction with care, and costs.

DETAILED DESCRIPTION:
Currently, over 80% of the population is expected to die of chronic life-limiting illnesses, predominant among which are the various manifestations of cardiovascular disease, cancer, dementia, and chronic lung disease. Patients with high cholesterol and those potentially at risk for atherosclerotic heart disease and stroke are often treated preventively with HMG Co-A reductase inhibitors (a.k.a., statins). Clinical trial evidence supports the use of statins for patients with hyperlipidemia and established ischemic heart disease to reduce risk of future cardiovascular events and mortality, and to reduce risk of future cardiovascular events in patients with multiple cardiac risk factors. Beneficial outcomes are evident in these trials after 3-6 years of treatment. Hence, statins are among the most prescribed medications in the world. In the United States, over 25% of Medicare beneficiaries take a statin medication. Statin medications are frequently continued until the patient can no longer eat or swallow at the end of life, because there are no evidence-based guidelines regarding when or how to discontinue medications for co-morbidities. The risks and costs vs. benefits of statins for palliative care patients, for whom prognosis is limited, remains a genuine clinical uncertainty. Meanwhile, medications for symptoms and other concerns accumulate as illness progresses, and therefore polypharmacy and compounding medication side effects are troublesome problems in the setting of advanced life-limiting illness. While multiple studies have demonstrated the benefit of long-term preventive statin use for patients at cardiovascular risk, other studies have supported the discontinuation of medications (specifically statins) in end-stage disease. A rational approach to medication discontinuation, specifically statin discontinuation, therefore has the potential to reduce patient burden, polypharmacy, and side effects, while also preserving healthcare resources for more beneficial interventions.

This study is a multi-site randomized controlled trial of discontinuing vs. continuing statin medications in patients with advanced life-limiting illness. Eligible participants are adults with advanced life-limiting illness with an estimated prognosis of 1-6 months who are on statins for primary or secondary prevention of cardiovascular events. The primary outcome is survival rate at 60 days; secondary outcomes address cardiovascular events, polypharmacy, medication adverse effects, quality of life (QOL), and measures of the patient's health-related experience. The primary hypothesis is that discontinuing statins will not influence survival. Secondary hypotheses are that discontinuation of statins will not adversely affect cardiovascular events or overall QOL, but will improve statin-related symptoms and decrease polypharmacy.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old;
* have an advanced life-limiting illness;
* have a life expectancy of >1 month, AND patient exhibits declining functional status, defined as a reduction in Australia-modified Karnofsky Performance Status (AKPS)22 score to <80% in the previous 3 months;
* be on a statin medication for primary or secondary prevention of cardiovascular disease for ≥3 months;
* have adequately intact cognitive status to provide informed consent and complete the baseline assessment, as evidenced by a Short Portable Mental Status Questionnaire (SPMSQ)23 score of ≥6;
* provide informed consent; and,
* speak and read English at or above a grade 5 level (per patient or caregiver report).

Exclusion Criteria:

* primary treating physician/care provider estimates their life expectancy as < 1 month;
* under the care of a primary treating physician/primary care provider who is unwilling to have the patient enrolled;
* not consenting;
* having known active cardiovascular disease or sufficient risk of active cardiovascular disease to require ongoing therapy with statin drugs, in the opinion of the treating physician; OR,
* exhibiting obvious symptoms of myositis, known liver function test (LFT) abnormalities of >2.5x the upper limit of normal (ULN), known creatine kinase (CK) abnormalities of >2.5x ULN, or other contraindications to continuing statins, in the opinion of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2011-06-03 (Actual); Primary Completion 2013-07-15 (Actual); Study Completion 2013-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Abernethy, MD, Principal Investigator — Duke University; Jean Kutner, MD, Principal Investigator — University of Colorado, Denver
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - San Diego Hospice and the Institute for Palliative Medicine, San Diego, California
  - University of Colorado, Denver, Denver, Colorado
  - Kaiser Permanente, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Four Seasons Hospice and Palliative Care, Flat Rock, North Carolina
  - Hospice of Western Reserve, Cleveland, Ohio
  - Capital Caring, Falls Church, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNeil MJ, Kamal AH, Kutner JS, Ritchie CS, Abernethy AP. The Burden of Polypharmacy in Patients Near the End of Life. J Pain Symptom Manage. 2016 Feb;51(2):178-83.e2. doi: 10.1016/j.jpainsymman.2015.09.003. Epub 2015 Sep 30. PMID 26432571
- [Background] Tjia J, Kutner JS, Ritchie CS, Blatchford PJ, Bennett Kendrick RE, Prince-Paul M, Somers TJ, McPherson ML, Sloan JA, Abernethy AP, Furuno JP. Perceptions of Statin Discontinuation among Patients with Life-Limiting Illness. J Palliat Med. 2017 Oct;20(10):1098-1103. doi: 10.1089/jpm.2016.0489. Epub 2017 May 18. PMID 28520522
- [Background] Portz JD, Kutner JS, Blatchford PJ, Ritchie CS. High Symptom Burden and Low Functional Status in the Setting of Multimorbidity. J Am Geriatr Soc. 2017 Oct;65(10):2285-2289. doi: 10.1111/jgs.15045. Epub 2017 Aug 30. PMID 28857119
- [Background] Hochman MJ, Kamal AH, Wolf SP, Samsa GP, Currow DC, Abernethy AP, LeBlanc TW. Anticholinergic Drug Burden in Noncancer Versus Cancer Patients Near the End of Life. J Pain Symptom Manage. 2016 Nov;52(5):737-743.e3. doi: 10.1016/j.jpainsymman.2016.03.020. Epub 2016 Sep 20. PMID 27663186
- [Result] Kutner JS, Blatchford PJ, Taylor DH Jr, Ritchie CS, Bull JH, Fairclough DL, Hanson LC, LeBlanc TW, Samsa GP, Wolf S, Aziz NM, Currow DC, Ferrell B, Wagner-Johnston N, Zafar SY, Cleary JF, Dev S, Goode PS, Kamal AH, Kassner C, Kvale EA, McCallum JG, Ogunseitan AB, Pantilat SZ, Portenoy RK, Prince-Paul M, Sloan JA, Swetz KM, Von Gunten CF, Abernethy AP. Safety and benefit of discontinuing statin therapy in the setting of advanced, life-limiting illness: a randomized clinical trial. JAMA Intern Med. 2015 May;175(5):691-700. doi: 10.1001/jamainternmed.2015.0289. PMID 25798575
- [Derived] Murali KP, Merriman JD, Yu G, Vorderstrasse A, Kelley AS, Brody AA. Complex Care Needs at the End of Life for Seriously Ill Adults With Multiple Chronic Conditions. J Hosp Palliat Nurs. 2023 Jun 1;25(3):146-155. doi: 10.1097/NJH.0000000000000946. Epub 2023 Apr 11. PMID 37040386
- [Derived] Murali KP, Yu G, Merriman JD, Vorderstrasse A, Kelley AS, Brody AA. Multiple Chronic Conditions among Seriously Ill Adults Receiving Palliative Care. West J Nurs Res. 2023 Jan;45(1):14-24. doi: 10.1177/01939459211041174. Epub 2021 Aug 25. PMID 34433344
- [Derived] Murali KP, Yu G, Merriman JD, Vorderstrasse A, Kelley AS, Brody AA. Latent Class Analysis of Symptom Burden Among Seriously Ill Adults at the End of Life. Nurs Res. 2021 Nov-Dec 01;70(6):443-454. doi: 10.1097/NNR.0000000000000549. PMID 34393192
- [Derived] Schenker Y, Park SY, Jeong K, Pruskowski J, Kavalieratos D, Resick J, Abernethy A, Kutner JS. Associations Between Polypharmacy, Symptom Burden, and Quality of Life in Patients with Advanced, Life-Limiting Illness. J Gen Intern Med. 2019 Apr;34(4):559-566. doi: 10.1007/s11606-019-04837-7. Epub 2019 Feb 4. PMID 30719645

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continue Statins | Discontinue Statins
Started | 192 | 189
Completed | 189 | 182
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Population: This was a 15-site, parallel-group, unblinded, pragmatic clinical trial. Eligibility included adults with an estimated life expectancy of between 1 month and 1 year, statin therapy for 3 months or more for primary or secondary prevention of cardiovascular disease and no recent active cardiovascular disease.
Groups:
- Continue Statins: Patients in the continuation group continued to receive statins.
- Discontinue Statins: Statin therapy was withdrawn from eligible patients who were randomized to the discontinuation group.
- Total: Total of all reporting groups
Arm/Group | Continue Statins | Discontinue Statins | Total
Number analyzed (Participants) | 192 | 189 | 381
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 35 | 73
  >=65 years | 154 | 154 | 308
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.5 (11.5) | 74.8 (11.7) | 74.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 91 | 171
  Male | 112 | 98 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 182 | 183 | 365
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 22 | 32 | 54
  White | 162 | 153 | 315
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 192 | 189 | 381

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Deaths Within 60 Days of Enrollment.
Description: To determine, among patients with life-limiting illness, if there is a difference in the proportion who die within 60 days after enrollment between patients for whom statins are discontinued vs. patients who are maintained on the medication.
Time Frame: Within 60 days of Subject Enrollment
Population: Intent to treat
Measure: Number (90% Confidence Interval); unit: proportion of deaths
Arm/Group | Continue Statins | Discontinue Statins
Number analyzed (Participants) | 192 | 189
proportion of deaths | 0.203 [0.156 to 0.257] | 0.238 [0.188 to 0.295]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Continue Statins | Discontinue Statins
All-Cause Mortality (participants affected / at risk) | 39/192 | 45/189
Serious Adverse Events (participants affected / at risk) | 4/192 | 6/189
Other Adverse Events (participants affected / at risk) | 4/192 | 7/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continue Statins (N=192) | Discontinue Statins (N=189)
Suicidal Ideation and severe depression (Psychiatric disorders) | 0 (0) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 0 (0) | 1 (1)
Shortness of Breath (General disorders) | 0 (0) | 3 (3)
Fever (General disorders) | 1 (1) | 0 (0)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Low Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rectal Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continue Statins (N=192) | Discontinue Statins (N=189)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Encephalpathy (Nervous system disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 1 (1) | 6 (6)
Fever (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rehospitalization (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Psychological Distress (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No